CLINICAL TRIAL: NCT05027737
Title: Early Ileostomy Closure Following Restorative Proctectomy for Rectal Cancer Patients: A North American Multicenter Randomized-Controlled Trial (RCT)
Brief Title: Early Ileostomy Closure for Rectal Cancer Patients in North America
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Associate Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-05-2022-2953
Record Dates: First submitted 2021-08-10; First posted 2021-08-30 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Ileostomy - Stoma; Rectal Cancer
Keywords: Early ileostomy closure; Comprehensive complication index; Bowel function; Quality of life; Recovery; Cost
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Multi-centre, assessor-blind, parallel-groups (1:1), pragmatic, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Ileostomy Closure (Experimental): Following a negative leak test (CT scan with rectally-administered water-soluble contrast on post-operative day 7, 8 or 9), patients will undergo standardized reversal of their diverting loop ileostomy (stapled side-side functional end-to end anastomosis, purse-string closure of the ileostomy wound, and no use of epidural analgesia) between post-operative days 10-14.
  Interventions: Procedure: Early Ileostomy Closure
- Traditional closure (control) (No Intervention): Following a negative leak test (CT scan with rectally-administered water-soluble contrast on post-operative day 7, 8 or 9), patients will undergo a standardized reversal of their diverting loop ileostomy. The latter will be performed with a stapled side-side functional end-to end anastomosis, purse-string closure of the ileostomy wound, and no use of epidural analgesia and will be performed no earlier than 12 weeks following their index surgery.

INTERVENTIONS:
Procedure: Early Ileostomy Closure — Following a negative leak test (CT scan with rectally-administered water-soluble contrast on post-operative day 7, 8 or 9), patients will undergo standardized reversal of their diverting loop ileostomy (stapled side-side functional end-to end anastomosis, purse-string closure of the ileostomy wound, and no use of epidural analgesia) between post-operative days 10-14.
  Arms: Early Ileostomy Closure

SUMMARY:
Our preliminary work demonstrates that there is buy-in from both patients and surgeons with regards to early ileostomy closure (EIC) for select rectal cancer patients undergoing restorative proctectomy (RP) and diverting loop ileostomy (DLI). The feedback from leaders in Europe further supports the need for a large scale randomized-controlled trial (RCT) on this subject in North America. Should the results of such a study be favourable, we believe it could support a change in practice that would be beneficial to patients and the health care system alike. Furthermore, our work will help identify which patients and practices are suitable for EIC.

The goal of our project is to determine whether EIC in rectal cancer patients undergoing RP with a DLI is safe, feasible and beneficial in a North American population. Specifically, our primary objective is to compare the severity of complications between patients undergoing EIC versus traditional (late) closure. Our secondary objectives include assessing the difference in quality of life (QoL), early and late bowel function, and cost of care between these two groups.

DETAILED DESCRIPTION:
Eligible adults (≥18 years-old) from one a large colorectal surgery practice in Canada who (1) underwent RP with creation of a DLI for the treatment of rectal cancer and (2) have a negative anastomotic leak test on post-operative day 7-9 which will consist of a flexible sigmoidoscopy and CT scan with rectally-administered water soluble contrast. Patients will be excluded if there is (1) peri-operative immunosuppression, (2) age-adjusted Charlson Comorbidity Index >6, (3) other major surgery during the index operation, and (4) any major complications (Clavien Dindo Grade III-V) following RP. Eligible participants will be randomized (1:1): Intervention group (EIC): Following a negative leak test, patients will undergo standardized reversal of their DLI (stapled side-side functional end-to end anastomosis, purse-string closure of the ileostomy wound and no use of epidural analgesia) between post-operative days 10-14. Control group (standard practice): Following a negative leak test, patients will undergo a standardized reversal of their DLI no earlier than 12 weeks following their index surgery.

The primary outcome will be comprehensive complication index (CCI) at 12 months following RP. Secondary outcomes will include: CCI at 2-, 6-, and 9-months following RP; recovery from surgery using the PROMIS 29 profile at 7- and 14-days post RP; bowel function, as measured using the Low Anterior Resection Syndrome (LARS) Score at 2-, 6-, 9-, and 12-months post-DLI closure; post-operative ileus, as defined by intolerance to oral intake in the absence of clinical or radiological signs of obstruction, will be measured prospectively after DLI closure; overall QoL, as measured by the EORTC CR30 and QLQ-CR38 at 0-, 2-, 6-, 9-, and 12-months post-RP; cost, as measured from the perspective of the healthcare system [length of hospital stay (RP, ileostomy closure, and any readmissions), interventions in any setting following RP, and appliance-related costs] will be assessed at 6- and 12-months post-index surgery. Treatment effect on the primary outcome (CCI at 12 months) will be modeled using linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years-old) patients
* Underwent restorative proctectomy by a laparoscopic, robotic, transanal total mesorectal excision, or open approach with creation of a diverting loop ileostomy for the treatment of rectal cancer
* Negative anastomotic "leak test" via CT scan with rectally-administered water-soluble contrast on post-operative day 7, 8 or 9.

Exclusion Criteria:

* Peri-operative immunosuppression (within 6 weeks of surgery date);
* Age-adjusted Charlson Comorbidity Index >6;
* Other major surgery during the index operation;
* Any major complications (Clavien Dindo Grade III or greater) following restorative proctectomy;
* Inability to speak or comprehend English or French and inability to give informed consent.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Complications | 12-months post-restorative proctectomy
  Comprehensive complication index

SECONDARY OUTCOMES:
Complications | 2-, 6-, and 9-months post-restorative proctectomy
  Comprehensive complication index
Occurrence of post-operative ileus following ileostomy reversal | Monitored for from date of ileostomy closure to day of discharge from hospital
  Intolerance to oral intake in the absence of clinical or radiological signs of obstruction, measured prospectively after diverting loop ileostomy closure
Cost of patient care (in dollars) | Calculated at 6- and 12-months post restorative proctectomy
  Measured from the perspective of the healthcare system, by combining cost of each hospital admission (restorative proctectomy, diverting loop ileostomy closure, and any readmissions), interventions in any setting following restorative proctectomy, and stoma appliance-related costs (measured based on the average number of bags and stoma appliances used per week by each patient).
Time to chemotherapy (weeks) | Starting from restorative proctectomy post-operative day 1 through the course of the study (1 year follow-up)
  Number of weeks elapsed from date of restorative proctectomy to date of initiation of adjuvant chemotherapy
Post-operative recovery | 1- and 2-weeks post-restorative proctectomy and diverting loop ileostomy as well as 30 days post-diverting loop ileostomy closure
  PROMIS-29 profile v2.0. PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation of that population. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Bowel function | 2-, 6-, 9-, and 12-months post-diverting loop ileostomy closure
  Low Anterior Resection Syndrome (LARS) Score. The score ranges from 0-42 with a score of 0-20 representing "No LARS", a score of 21-29 representing "Minor LARS" and a score of 30-42 representing "Major LARS".
EORTC QLQ-C30 score | Baseline (day of patient recruitment), 2-, 6-, 9-, and 12-months post-restorative proctectomy
  Health-related quality of life of cancer patients. All of the scale ranges in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
EORTC QLQ-CR29 score | Baseline (day of patient recruitment), 2-, 6-, 9-, and 12-months post-restorative proctectomy
  Health-related quality of life of colorectal cancer patients. All of the scale ranges in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec